CLINICAL TRIAL: NCT05611320
Title: Assessing and Amplifying Parent Support for Locally Sourced Produce in Barbados
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inter-American Development Bank (Other)
Collaborators: Busara Center for Behavioral Economics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-BA-1
Record Dates: First submitted 2022-10-19; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Nutrition Poor
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awareness Campaign (Experimental): Raise awareness among parents about how and why to use local produce in their kid's meals.
  Interventions: Other: Awareness campaign - communications campaign
- Online Shopping (Experimental): Provide information about an online shopping platform where the parents can shop for local produce online, and have it delivered, to disrupt their current ingredient-selection habits.
  Interventions: Other: Online shopping

INTERVENTIONS:
Other: Awareness campaign - communications campaign — How this concept would work in a full deployment:
  1. Develop a set of images of healthy meals with local produce. The meals will be child-friendly and easy to prepare.
  2. Develop educational content to accompany the images, on the importance of shopping for local produce, and seasonality (when to use what). Optionally work with farmer associations to inform the seasonal options.
  3. Package the materials as posters and/or digital infographics. The materials include a link to the campaign website, which has more information about nutrition, local produce and recipes to inspire parents.
  4. Partner with government agencies (e.g., ministry of health) to deploy the posters in local supermarkets, and in newspapers and on social media. Make the materials available to the farmer associations for their dissemination as well.
  Arms: Awareness Campaign
Other: Online shopping — Provide information on an online shopping site where the parents can shop for local produce online, and have it delivered to their homes, to disrupt their current ingredient-selection habits. Working backwards from a potential broad implementation, here we identify key risks along the path, and examine how to use the pilot to de-risk those areas.
  Arms: Online Shopping

SUMMARY:
This study seeks to promote consumption of locally sourced foods among school going children in Barbados. The study targets parents/care givers of school going children aged 18 years and below. Parents have been chosen as the target for this study because they shape the meals that their children consume through two primary routes; a) direct purchase of meal ingredients and b) political influence on school based meal programs. The study seeks to achieve this by first identifying the behavioral obstacles for consumption of locally sourced produce through exploratory and desk research and then designing interventions to address the obstacles.

DETAILED DESCRIPTION:
This study will be rolled out as a digital interface experiment where the survey and intervention prompts will be programmed on OTree platform with pre-randomized assignments of the participants into either treatment or control groups. Busara Center for Behavioral Economics has partnered with a local organization named FutureBarbados who are part of the Government of Barbados. The organization will avail census data for parents with school going children below 18 years of age in Barbados. Busara will then randomly sample a pool of 1500 parents who will be sent a link to the programmed survey and intervention prompts to fill out. The process will entail first a consenting process which will be displayed on their phone screens upon opening the link. The consent information will outline clearly the purpose of their study, the length of the survey, data confidentiality, the voluntary nature of participation as well as contact information in the event they would like further clarification before making the decision to take part in the study.

Once the participants consent to take part in the study the survey will have been programmed to assign them the respective survey depending on the treatment or control assignment.

The assignments are as follows:

* Control group 1: This will involve the provision of innocuous information about food. This provides a control group that is similar to the treatment groups in terms of the amount of time and cognitive effort demanded from them. This allows for a baseline measurement of parental interest in local produce.
* Control group 2: This will involve provision of general, positive information about the use of local produce in school meals. This is a secondary control that allows for the separate estimation of the effect of increasing attention to local produce, and serves to control for demand effects of the experiment itself.
* Treatment group 1: This will include an awareness campaign designed for parents. The campaign will consist of a series of photos of healthy meals showcasing how to use local produce. The meals will be child-friendly and easy to prepare. The messaging on the campaign will include educational content on 1) the importance of shopping for local produce to support farmers and the local community rather than relying solely on imported produce. 2) Seasonality of local produce; when to use what? This is intended to support parents to plan their meals according to availability of certain local produce with the ultimate aim of obtaining a healthy diet affordably
* Treatment group 2: This will provide information promoting of an online market platform where one can order local produce to be delivered directly to their homes.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of school going children aged 18 years and below and living in Barbados
* Parents/Caregivers of school going children aged 18 years and below who have access to a mobile phone

Exclusion Criteria:

- Parents /caregivers whose children are above 18 years old, do not live in Barbados and do not have access to a mobile phone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Voucher Selection | Through study completion, an average of 1 year
  Knowledge, attitudes and political support for local food, as well as a final measure of whether the respondent would rather receive a voucher for a store that sells local produce or a voucher for a store that sells imported food.
  Parents will be incentivized for their participation in the study with 10 Bajan Dollars for the purchase of food, and will be entered into a sweepstakes for 2000 Bajan Dollars (1,000 USD). At the end of the intervention given above, they are asked whether they would like a voucher for either:
  1. A fast food restaurant
  2. A local produce market
  The voucher selection is an incentive-compatible proxy for purchasing local produce or imported goods. This choice is made in full awareness of the frictions that parents face to sourcing produce from farmers markets, versus the ease of a supermarket: the study measures the impact of the interventions on behavior change in their real context, not in a hypothetical, friction-free choice environment.
Political support for prioritization of local food | Through study completion, an average of 1 year
  Parents will be asked to rank order their preference for government policies among numerous (real) options -from job creation programs to climate change; embedded in that list will be a program for locally sourced produce for kids. Each arm's average ranking for the local produce option serves as the political support outcome measure.